CLINICAL TRIAL: NCT02376465
Title: A Pilot Evaluation of an Experimental BLI4600 Formulation for Bowel Preparation in Adult Patients Undergoing Colonoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BLI4600-201
Record Dates: First submitted 2015-02-26; First posted 2015-03-03 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Bowel Preparation for Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BLI4600 Regimen 1 (Experimental): Oral bowel preparation for colonoscopy
  Interventions: Drug: BLI4600 bowel preparation
- BLI4600 Regimen 2 (Experimental): Oral bowel preparation for colonoscopy
  Interventions: Drug: BLI4600 bowel preparation
- PEG based below preparation (Active Comparator): Oral bowel preparation for colonoscopy
  Interventions: Drug: PEG based bowel preparation

INTERVENTIONS:
Drug: BLI4600 bowel preparation — Oral bowel preparation for colonoscopy
  Arms: BLI4600 Regimen 1; BLI4600 Regimen 2
Drug: PEG based bowel preparation — Oral bowel preparation for colonoscopy
  Arms: PEG based below preparation

SUMMARY:
To evaluate the safety, tolerance and efficacy of BLI4600 in multiple dosing regimens as a bowel preparation prior to colonoscopy in adult patients.

ELIGIBILITY:
Inclusion Criteria:

Male or female outpatients who are undergoing colonoscopy for a routinely accepted indication

At least 18 years of age

If female, and of child-bearing potential, is using an acceptable form of birth control (hormonal birth control, IUD, double-barrier method, depot contraceptive, abstinent, or vasectomized spouse).

Negative urine pregnancy test at screening, if applicable

In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Exclusion Criteria:

Subjects with known or suspected ileus, severe ulcerative colitis, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis or megacolon.

Subjects who had previous significant gastrointestinal surgeries (e.g. colostomy, colectomy, gastric bypass, stomach stapling).

Subjects with uncontrolled pre-existing electrolyte abnormalities, such as hypernatremia, hyponatremia, hyperphosphatemia, hypokalemia, hypocalcemia, dehydration, or those secondary to the use of diuretics or angiotensin converting enzyme (ACE) inhibitors.

Subjects with a prior history of renal, liver or cardiac insufficiency.

Subjects with impaired consciousness that predisposes them to pulmonary aspiration.

Subjects undergoing colonoscopy for foreign body removal and/or decompression.

Subjects who are pregnant or lactating, or intending to become pregnant during the study.

Subjects of childbearing potential who refuse a pregnancy test.

Subjects allergic to any preparation components.

Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures.

Subjects who have participated in an investigational surgical, drug, or device study within the past 30 days.

Subjects who withdraw consent before completion of Visit 1 procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
% of subjects with successful preparation on a 4 point scale (1 = poor, 2 = fair, 3 = good, 4 = excellent) | 1 Day
  % of subjects with successful preparation by colonoscopist on a 4 point scale (1 = poor, 2 = fair, 3 = good, 4 = excellent)

SECONDARY OUTCOMES:
Ottawa Bowel Preparation Scale Score | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, MPH, Study Director — Braintree Laboratories, Inc.
Locations (1):
- University of South Alabama, Mobile, Alabama, United States